CLINICAL TRIAL: NCT00571428
Title: Modified-blind, Randomized, Multicenter, Single Dose, Two-way Crossover Study of Arformoterol Tartrate Inhalation Solution 15 Micrograms Twice A Day Versus 30 Micrograms Once A Day in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy Safety Study of Arformoterol QD Dosing Versus BID Dosing in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 091-903
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2009-07-02 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Bronchitis; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 15 mcg BID / 30 mcg QD (Experimental): Arformoterol 15 microgram twice a day (BID) taken each morning and evening for one visit followed by Arformoterol 30 microgram once a day (QD) in the morning and placebo in the evening for the next visit.
  Interventions: Drug: Arformoterol Tartrate Inhalation Solution; Drug: Placebo
- 30 mcg QD / 15 mcg BID (Experimental): Arformoterol 30 microgram once a day (QD) in the morning and placebo in the evening for one visit followed by Arformoterol 15 microgram twice a day (BID) in the morning and evening for the next visit.
  Interventions: Drug: Arformoterol Tartrate Inhalation Solution; Drug: Placebo

INTERVENTIONS:
Drug: Arformoterol Tartrate Inhalation Solution — Nebulized arformoterol tartrate inhalation solution 15 microgram twice a day (BID)
  Other Names: Brovana
Drug: Arformoterol Tartrate Inhalation Solution — Nebulized arformoterol tartrate inhalation solution 30 microgram once a day (QD)
  Other Names: Brovana
Drug: Placebo — Placebo inhalation solution (citrate buffered 0.9% saline solution) once a day

SUMMARY:
To evaluate the efficacy and safety of arformoterol tartrate inhalation solution 30μg/4mL QD (two 15μg/2mL dosed in combination) over a 24-hour period compared to arformoterol tartrate inhalation solution 15μg/2 mL BID in subjects with COPD.

DETAILED DESCRIPTION:
This is a modified blind, randomized, multicenter, single dose two-way crossover study to assess the efficacy and safety of arformoterol 15μg BID versus arformoterol 30μg QD in subjects with COPD. Subject participation will last approximately three weeks and will include a screening visit, two 24-hour visits, and a follow up telephone call. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be at least 45 years old at the time of consent.
* Subjects must have a pre-established primary clinical diagnosis of COPD.
* Subjects must have a baseline FEV1 of ≤ 65% of predicted normal value at Visit 1.
* Subjects must have a FEV1 ≥ 0.70L at Visit 1.
* Subjects must have a FEV1/forced vital capacity (FVC) ratio of ≤ 70% at Visit 1.

Exclusion Criteria:

* Subjects who do not have a 15 pack-year smoking history and a baseline breathlessness severity grade of 2 (as measured by the Modified Medical Research Council [MMRC] Dyspnea Scale Score) at Screening.
* Subjects with life-threatening/unstable respiratory status, including upper or lower respiratory tract infection, within the previous 30 days prior to Visit

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pulmonary Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (4):
- United States (4):
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Spartanburg, South Carolina

REFERENCES:
- [Derived] Panettieri RA Jr, MacIntyre N, Sims M, Kerwin E, Fogarty C, Noonan M, Claus R, Andrews WT. Comparison of the efficacy and safety of arformoterol 15 microg twice daily and arformoterol 30 microg once daily in COPD: a single-dose, multicenter, randomized, modified-blind, two-way crossover study. Clin Ther. 2009 Aug;31(8):1716-23. doi: 10.1016/j.clinthera.2009.08.012. PMID 19808130

RESULTS

PARTICIPANT FLOW:
Groups:
- 15 Mcg BID / 30 Mcg QD: Arformoterol 15 mcg twice a day (morning and evening) for one visit followed by Arformoterol 30 mcg once a day (morning) and placebo (evening) for the next visit.
- 30 Mcg QD / 15 Mcg BID: Arformoterol 30 mcg once a day (morning) and placebo (evening) for one visit followed by Arformoterol 15 mcg twice a day (morning and evening) for the next visit.
Period: Overall Study
Arm/Group | 15 Mcg BID / 30 Mcg QD | 30 Mcg QD / 15 Mcg BID
Started | 15 | 18
Completed | 15 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 Mcg BID / 30 Mcg QD | 30 Mcg QD / 15 Mcg BID | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 7 | 7 | 14.0
  >=65 years | 8 | 11 | 19.0
Age Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (9.3) | 64.9 (8.7) | 64.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13.0
  Male | 9 | 11 | 20.0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0.0
  Asian | 0 | 0 | 0.0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0.0
  Black or African American | 2 | 2 | 4.0
  White | 13 | 16 | 29.0
  More than one race | 0 | 0 | 0.0
  Unknown or Not Reported | 0 | 0 | 0.0
Inhaled Corticosteroid Use at Baseline [Number; unit: participants] — This measure answers the question: Does the patient use a corticosteroid inhaler at the baseline visit?
  participants
    Yes | 1 | 4 | 5.0
    No | 14 | 14 | 28.0
Participants Categorized by the Number of Pack Years Smoked [Number; unit: participants] — Pack years smoked is a way to measure the amount a person has smoked over a long period of time. It is calculated by taking the number of cigarettes smoked per day times the the number of years smoked divided by 20 (cigarettes per pack).
  participants
    >=15 years - <25 years | 1 | 2 | 3.0
    >=25 years - < 30 years | 0 | 3 | 3.0
    >=30 years | 14 | 13 | 27.0
Participants Categorized by the Number of Packs Currently Smoked per Day [Number; unit: participants] — This measure gives an indication of the quantity of cigarettes currently smoked per day.
  participants
    >0 -1 pack | 5 | 4 | 9.0
    >1 -2 packs | 3 | 3 | 6.0
    >2 - 4 packs | 0 | 0 | 0.0
    > 4 packs | 0 | 0 | 0.0
    Currently does not smoke | 7 | 11 | 18.0

OUTCOME MEASURES:

1. Primary Outcome: Time-Normalized Area Under the Change From Pre-Dose Curve for Forced Expiratory Volume in One Second Measured Over 24 Hours
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome measures the change from pre-dose for a series of FEV1 readings taken within 24 hours of dosing.
Time Frame: 0-24 hours post dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: liters
Groups:
- 15 Mcg BID: Arformoterol 15 mcg twice a day (morning and evening)
- 30 Mcg QD: Arformoterol 30 mcg once a day (morning) and placebo (evening)
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 32 | 32
liters | 0.156 (0.156) | 0.173 (0.183)
Statistical Analysis 1: Comparison: 15 Mcg BID vs 30 Mcg QD; Test type: Non-Inferiority or Equivalence — Equivalence was defined a priori such that 90%CI for the difference between therapies had to fall entirely within +/- 0.07L; Mixed Models Analysis; Treatment group, treatment sequence, predose FEV1, & Visit number are fixed effects; subject within treatment sequence is a random effect; Mean Difference (Final Values) = 0.011, 90% CI [-0.015 to 0.037]

2. Secondary Outcome: Time-Normalized Area Under the Change From Pre-Dose Curve for Forced Expiratory Volume in One Second Measured Over 12 Hours
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome measures the change from pre-dose for a series of FEV1 readings taken within 12 hours of dosing.
Time Frame: 0-12 hours
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 32 | 32
liters | 0.148 (0.152) | 0.214 (0.163)
Statistical Analysis 1: Comparison: 15 Mcg BID vs 30 Mcg QD; Test type: Non-Inferiority or Equivalence — Equivalence was defined a priori such that 90%CI for the difference between therapies has to fall entirely within +/- 0.07L; Mixed Models Analysis; Treatment group, treatment sequence, pre-dose FEV1, & Visit Number are fixed effects; subjects within treatment sequence is a random effect; Mean Difference (Final Values) = 0.062, 90% CI [0.035 to 0.090]

3. Secondary Outcome: Time-Normalized Area Under the Change From Pre-Dose Curve for Forced Expiratory Volume in One Second Measured Between 12-24 Hours
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome measures the change from pre-dose for a series of FEV1 readings taken between 12 and 24 hours of dosing.
Time Frame: 12-24 hours
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 30 | 32
liters | 0.179 (0.154) | 0.132 (0.211)
Statistical Analysis 1: Comparison: 15 Mcg BID vs 30 Mcg QD; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Median Difference (Final Values) = -0.035, 90% CI [-0.079 to 0.008]

4. Secondary Outcome: Change in Forced Expiratory Volume in One Second From Pre-dose to the 24 Hour Time Point
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome measures the change in FEV1 from pre-dose to the readings taken 24 hours post-dose, which represents the trough in dose level.
Time Frame: pre-dose and 24 hours post-dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 31 | 31
liters | 0.144 (0.161) | 0.120 (0.195)
Statistical Analysis 1: Comparison: 15 Mcg BID vs 30 Mcg QD; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Median Difference (Final Values) = -0.030, 90% CI [-0.086 to 0.026]

5. Secondary Outcome: Forced Expiratory Volume in One Second Measurements Pre-dose and at Each Assessed Time Point Post-dose
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome offers the FEV1 readings taken pre-dose and at various time points within 24 hours post-dose.
Time Frame: pre-dose, immediately post-dose, 30 min, 1,2,4,6,8,10,12, 12.5,13,14,16,23,24 hours post first dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 33 | 33
liters
  Pre-dose (n=32,32) | 1.184 (0.366) | 1.179 (0.342)
  Immediately post first dose (n=32,33) | 1.332 (0.418) | 1.358 (0.386)
  30 minutes (n=33,33) | 1.349 (0.392) | 1.384 (0.374)
  1 hour post first dose (n=33,33) | 1.362 (0.387) | 1.401 (0.394)
  2 hours post first dose (n=33,33) | 1.378 (0.375) | 1.419 (0.378)
  4 hours post first dose (n=33,33) | 1.342 (0.374) | 1.429 (0.375)
  6 hours post first dose (n=32,30) | 1.359 (0.426) | 1.414 (0.384)
  8 hours post first dose (n=32,30) | 1.303 (0.402) | 1.373 (0.397)
  10 hours post first dose (n=31,30) | 1.308 (0.371) | 1.371 (0.411)
  12 hours post first dose (n=30,32) | 1.270 (0.365) | 1.327 (0.400)
  12.5 hours post first dose (n=30,32) | 1.359 (0.359) | 1.332 (0.409)
  13 hours post first dose (n=30,32) | 1.389 (0.375) | 1.330 (0.378)
  14 hours post first dose (n=30,32) | 1.397 (0.389) | 1.337 (0.411)
  16 hours post first dose (n=32,33) | 1.368 (0.357) | 1.344 (0.420)
  23 hours post first dose (n=30,32) | 1.297 (0.373) | 1.252 (0.412)
  24 hours post first dose (n=31,32) | 1.296 (0.363) | 1.279 (0.417)

6. Secondary Outcome: Change in Forced Expiratory Volume in One Second From Pre-dose To Each Assessed Time Point Post-Dose
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome offers the change in FEV1 readings between pre-dose and various time points within 24 hours post-dose.
Time Frame: Immediately post first dose, 30 min, 1,2,4,6,8,10,12,12.5,13,14,16,23,24 hours post first dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 33 | 33
liters
  Immediately post first dose (n=32,32) | 0.148 (0.109) | 0.187 (0.137)
  30 minutes post first dose (n=32,32) | 0.168 (0.128) | 0.211 (0.157)
  1 hour post first dose (n=32,32) | 0.179 (0.131) | 0.229 (0.156)
  2 hours post first dose (n=32,32) | 0.193 (0.141) | 0.243 (0.160)
  4 hours post first dose (n=32,32) | 0.161 (0.155) | 0.248 (0.172)
  6 hours post first dose (n=32,30) | 0.175 (0.182) | 0.243 (0.181)
  8 hours post first dose (n=32,30) | 0.119 (0.199) | 0.202 (0.191)
  10 hours post first dose (n=30,30) | 0.145 (0.165) | 0.200 (0.203)
  12 hours post first dose (n=30,32) | 0.105 (0.167) | 0.148 (0.197)
  12.5 hours post first dose (n=30,32) | 0.193 (0.152) | 0.153 (0.211)
  13 hours post first dose (n=30,32) | 0.223 (0.148) | 0.151 (0.198)
  14 hours post first dose (n=30,32) | 0.232 (0.175) | 0.158 (0.229)
  16 hours post first dose (32,32) | 0.184 (0.178) | 0.163 (0.237)
  23 hours post first dose (n=30,31) | 0.132 (0.189) | 0.088 (0.211)
  24 hours post first dose (n=31,31) | 0.144 (0.161) | 0.120 (0.195)

7. Secondary Outcome: Percent of Predicted Forced Expiratory Volume at One Second at Pre-dose and Each Assessed Time Point Post-Dose
Description: Predicted FEV1 is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. This outcome uses actual FEV1 readings to generate the percent of the estimated healthy lung function at specified time points.
Time Frame: Pre-dose, Immediately post first dose, 30 min, 1,2,4,6,8,10,12,12.5,13,14,16,23,24 hours post first dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Percent of Predicted FEV1
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 33 | 33
Percent of Predicted FEV1
  Pre-dose (n=32,32) | 40.717 (10.522) | 40.784 (10.554)
  Immediately post first dose (n=32,33) | 45.504 (10.938) | 46.396 (10.617)
  30 min post first dose (n=33,33) | 45.990 (10.407) | 47.303 (10.250)
  1 hour post first dose (n=33,33) | 46.456 (10.638) | 47.816 (10.469)
  2 hours post first dose (n=33,33) | 47.136 (10.393) | 48.559 (10.352)
  4 hours post first dose (n=33,33) | 45.839 (10.366) | 48.832 (9.868)
  6 hours post first dose (n=32,30) | 46.294 (10.678) | 48.133 (10.958)
  8 hours post first dose (n=32,30) | 44.534 (10.892) | 46.491 (10.507)
  10 hours post first dose (n=31,30) | 44.913 (10.947) | 46.360 (10.932)
  12 hours post first dose (n=30,32) | 43.885 (10.726) | 45.446 (10.821)
  12.5 hours post dose (n=30,32) | 46.935 (10.728) | 45.560 (11.216)
  13 hours post first dose (n=30,32) | 47.848 (10.703) | 45.723 (11.043)
  14 hours post first dose (n=30,32) | 48.051 (10.730) | 45.711 (11.116)
  16 hours post first dose (n=32,33) | 46.977 (10.236) | 45.599 (11.074)
  23 hours post first dose (n=30,32) | 44.876 (11.561) | 42.793 (11.537)
  24 hours post first dose (n=31,32) | 44.844 (10.730) | 43.729 (11.178)

8. Secondary Outcome: Change in Percent of Predicted Forced Expiratory Volume at One Second (FEV1) at Each Assessed Time Point Post-Dose Compared to Pre-Dose
Description: Predicted FEV1 is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. This outcome uses actual FEV1 readings to generate the change in percent of the estimated healthy lung function at specified time points compared to the pre-dose value.
Time Frame: Immediately post first dose, 30 min, 1,2,4,6,8,10,12,12.5,13,14,16,23,24 hours post first dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: percent of predicted FEV1
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 33 | 33
percent of predicted FEV1
  Immediately post first dose (n=32,32) | 4.787 (3.274) | 6.028 (4.296)
  30 minutes post first dose (n=32,32) | 5.574 (3.880) | 6.917 (4.911)
  1 hour post first dose (n=32,32) | 5.980 (4.124) | 7.437 (4.578)
  2 hours post first dose (n=32,32) | 6.570 (4.607) | 8.055 (4.761)
  4 hours post first dose (n=32,32) | 5.399 (4.820) | 8.189 (5.103)
  6 hours post first dose (n=32,30) | 5.576 (5.237) | 7.904 (5.786)
  8 hours post first dose (n=32,30) | 3.816 (6.276) | 6.261 (6.101)
  10 hours post first dose (n=30,30) | 4.810 (5.710) | 6.130 (6.679)
  12 hours post first dose (n=30,32) | 3.507 (5.382) | 4.662 (6.733)
  12.5 hours post first dose (n=30,32) | 6.557 (5.216) | 4.776 (7.496)
  13 hours post first dose (n=30,32) | 7.470 (4.903) | 4.939 (6.978)
  14 hours post first dose (n=30,32) | 7.672 (5.398) | 4.927 (7.734)
  16 hours post first dose (n=32,32) | 6.259 (5.767) | 4.937 (8.080)
  23 hours post first dose (n=30,31) | 4.498 (6.276) | 2.457 (7.732)
  24 hours post first dose (n=31,31) | 4.875 (4.925) | 3.528 (6.540)

9. Secondary Outcome: Peak Percent of Predicted Forced Expiratory Volume at One Second (FEV1) Over 12 Hours Post-Dose.
Description: Predicted FEV1 is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. This outcome uses actual FEV1 readings to generate the percent of the estimated healthy lung function and reports the highest percent found within 12 hours of dosing.
Time Frame: 12 hours
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: percent of predicted FEV1
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 33 | 33
percent of predicted FEV1 | 49.399 (10.738) | 51.251 (10.606)
Statistical Analysis 1: Comparison: 15 Mcg BID vs 30 Mcg QD; Test type: Superiority or Other; Mixed Models Analysis; Treatment group, treatment sequence, pre-dose FEV1, & Visit number are fixed effects; subject within treatment sequence is a random effect; Mean Difference (Final Values) = 1.694, 90% CI [0.525 to 2.862]

10. Secondary Outcome: Peak Change in Forced Expiratory Volume at One Second (FEV1) Within 12 Hours Post Dose Compared to Pre-dose
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer. This outcome measures the change in FEV1 from pre-dose to the readings taken 12 hours post-dose, and reports the largest change during that time.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 32 | 32
liters | 0.269 (0.154) | 0.324 (0.166)
Statistical Analysis 1: Comparison: 15 Mcg BID vs 30 Mcg QD; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.052, 90% CI [0.015 to 0.090]

11. Secondary Outcome: Time to Onset of 15 Percent Response Within 12 Hours of Dosing
Description: Time to a 15 percent improvement in forced expiratory volume in one second (FEV1) within 12 hours of dosing. Only patients who achieved at least a 15 percent improvement are included.
Time Frame: 12 hours post first dose
Population: Intent to treat population. Limited to those patients who had a 15% response.
Measure: Median (Full Range); unit: minutes
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 20 | 25
minutes | 7.75 [1.26 to 111.28] | 2.43 [1.13 to 692.29]

12. Secondary Outcome: Time to Onset of Response of Both a 12 Percent Increase and 200 Milliliter Increase Within 12 Hours of Dosing
Description: Time to a 12 percent improvement in forced expiratory volume in one second (FEV1) AND a 200 milliliter increase in FEV1 within 12 hours of dosing. Only patients who met both conditions are included
Time Frame: up to 12 hours post dose
Population: Intent to treat population. Limited to patients who met both criteria: a 12 percent increase in FEV1 and a 200 milliliter increase in FEV1
Measure: Median (Full Range); unit: minutes
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 20 | 25
minutes | 12.62 [1.22 to 343.91] | 2.86 [1.22 to 595.60]

13. Secondary Outcome: Time to Onset of Response of Both a 12 Percent Increase and 200 Milliliter Increase in Forced Expiratory Volume in One Second Within 12 Hours of Dosing
Description: Forced vital capacity is the total amount of air that can forcibly be blown out after full inspiration.
Time Frame: pre-dose, immediately post first dose, 30 min, 1,2,4,6,8,10,12, 12.5, 13, 14, 16, 23,24 hours post first dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 33 | 33
minutes
  Pre-dose (n=32,32) | 2.545 (0.718) | 2.601 (0.746)
  Immediately post first dose (n=32,33) | 2.838 (0.790) | 2.905 (0.796)
  30 minutes post first dose (n=33,33) | 2.903 (0.814) | 2.953 (0.808)
  1 hour post first dose (n=33,33) | 2.918 (0.771) | 3.003 (0.846)
  2 hours post first dose (n=33,33) | 2.931 (0.804) | 3.030 (0.800)
  4 hours post first dose (n=33,33) | 2.871 (0.783) | 3.028 (0.849)
  6 hours post first dose (n=32,30) | 2.849 (0.822) | 2.993 (0.844)
  8 hours post first dose (n=32,30) | 2.776 (0.828) | 2.940 (0.850)
  10 hours post first dose (n=31,30) | 2.796 (0.852) | 2.906 (0.910)
  12 hours post first dose (n=30,32) | 2.702 (0.832) | 2.797 (0.862)
  12.5 hours post first dose (n=30,32) | 2.852 (0.832) | 2.796 (0.852)
  13 hours post first dose (n=30,32) | 2.905 (0.876) | 2.815 (0.829)
  14 hours post first dose (n=30,32) | 2.878 (0.839) | 2.813 (0.862)
  16 hours post first dose (n=32,33) | 2.854 (0.824) | 2.812 (0.869)
  23 hours post first dose (n=30,32) | 2.733 (0.834) | 2.700 (0.866)
  24 hours post first dose (n=31,32) | 2.774 (0.809) | 2.763 (0.875)

14. Secondary Outcome: Change in Forced Vital Capacity From Pre-dose to Each Post-Dose Assessed Time Point
Description: Forced vital capacity is the total amount of air that can forcibly be blown out after full inspiration. The measure compares the change from pre-dose reading to each post-dose time point.
Time Frame: immediately post first dose, 30 min, 1,2,4,6,8,10,12, 12.5, 13, 14, 16, 23,24 hours post first dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 15 Mcg BID | 30 Mcg QD
Number analyzed (Participants) | 33 | 33
liters
  Immediately post first dose (n=32,32) | 0.293 (0.240) | 0.290 (0.274)
  30 minutes post first dose (n=32,32) | 0.334 (0.264) | 0.340 (0.274)
  1 hour post first dose (n=32,32) | 0.352 (0.270) | 0.390 (0.310)
  2 hours post first dose (n=32,32) | 0.355 (0.277) | 0.411 (0.335)
  4 hours post first dose (n=32,32) | 0.296 (0.308) | 0.398 (0.369)
  6 hours post first dose (n=32,30) | 0.304 (0.331) | 0.384 (0.364)
  8 hours post first dose (n=32,30) | 0.231 (0.352) | 0.331 (0.393)
  10 hours post first dose (n=30,30) | 0.246 (0.345) | 0.297 (0.386)
  12 hours post first dose (n=30,32) | 0.175 (0.319) | 0.196 (0.359)
  12.5 hours post first dose (n=30,32) | 0.325 (0.348) | 0.195 (0.355)
  13 hours post first dose (n=30,32) | 0.378 (0.326) | 0.214 (0.359)
  14 hours post first dose (n=30,32) | 0.351 (0.374) | 0.213 (0.383)
  16 hours post first dose (n=32,32) | 0.308 (0.378) | 0.183 (0.414)
  23 hours post first dose (n=30,31) | 0.206 (0.348) | 0.088 (0.380)
  24 hours post first dose (n=31,31) | 0.257 (0.337) | 0.148 (0.344)

ADVERSE EVENTS:
Description: Total number of participants in study is 33. 33 particpants at risk in each treatment arm due to cross over study design.
Arm/Group | 15 Mcg BID | 30 Mcg QD
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 2/33 | 3/33
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 Mcg BID (N=33) | 30 Mcg QD (N=33)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Arthraglia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Single day/dose; small numbers of subjects; difference between arms (2mL vs 4mL per dose); Predefined +/-0.07L equivalence is arbitrarily lower than the clinically recognized 0.1L. Hence, clinical efficacy & safety conclusions are difficult to reach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the 60 to 180 day restriction above, since this is a multicenter study, first publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish